CLINICAL TRIAL: NCT03051594
Title: Reliability of Fluorescent Camera and Caries Detection Dye Versus the Visual Tactile Method in Determining Caries Excavation Endpoint Using Microbiological Assessment (Randomized Clinical Trial)
Brief Title: Reliability of Fluorescent Camera and Caries Detection Dye Versus the Visual Tactile Method
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohamed mohamed sabry mohamed, Resident at conservative department, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: oper 603
Record Dates: First submitted 2017-02-03; First posted 2017-02-13 (Actual); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The side to which interventions or control is assigned to will be recorded and all records of all patients will be kept with the main supervisor . The operator will not be blinded as the difference in application protocol of the restorative materials prohibited blinding of the operator; however, the patient, Statisticians and Outcome assessors will be blinded to the material assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- visual tactile assessment (Active Comparator): dentine sample collection and then bacterial count by Digital colony counter, Agar diffusion test after visual tactile assessment.
  Interventions: Diagnostic Test: visual tactile assessment
- caries detector dye (Active Comparator): dentine sample collection and then bacterial count by Digital colony counter, Agar diffusion test after after using caries detector dye to determine the excavation endpoint.
  Interventions: Other: caries detector dye
- fluorescent camera (Experimental): dentine sample collection and then bacterial count by Digital colony counter, Agar diffusion test after after using fluorescent camera to determine the excavation endpoint.
  Interventions: Device: fluorescent camera

INTERVENTIONS:
Device: fluorescent camera — used too detect residual caries depending on the bacterial byproducts.
  Arms: fluorescent camera
Other: caries detector dye — dye used to detect the residual caries.
  Arms: caries detector dye
Diagnostic Test: visual tactile assessment — method usually used to detect the residual caries.
  Arms: visual tactile assessment

SUMMARY:
1. Three dentinal carious lesions will be chosen in this study and will be in the same patient.
2. Using local anaesthesia and rubber dam, the operative field will disinfected with 1% hypochlorite, and the dentine lesions should be exposed with a high-speed diamond bur by removing covering enamel.
3. Before the excavation dentine samples are collected for baseline bacteriological assessment .
4. Excavation will be carried out using new slow speed round burs and hand excavators.
5. The excavation end point of one cavity will be determined using visual tactile method. The two other cavities will be inspected with fluorescent camera or caries detector dye (CDD) methods to determine excavation endpoint respectively.
6. After excavation, dentine samples from the three cavities will be collected using a sterile excavator for the bacteriological assessment.

   * Number of visits & follow up period: all procedures will be done at the same visit and there is no follow up period.

Direct benefit of the research to the human volunteer: to determine the excavation endpoint to ensure complete caries removal and prevent it's recurrence in the future.

Scientific value and social benefits: to reach the best method to determine the excavation endpoint.

Expected risk to the human subjects: the ordinary side effects associated with any restorative treatment and no of the study variable has side effect on the patient and in case of any side effect due to the restorative treatment, the participant will directly contact the operator.

DETAILED DESCRIPTION:
II.1. Study setting

This clinical study will be held in the Clinic of Conservative Dentistry Department, Faculty of Oral and Dental Medicine, Cairo University, Egypt. The researcher will bear ultimate responsibility for all activities associated with the conduct of a research project including recruitment of patients , explaining and performing the procedures to them.

II.2. Variables of the study:

A total of 20 patients will participate in the study. Each patient will have 3 carious teeth. Resulting in a total of 60 carious lesions.

II.3. Trial Description:

II.3.a excavation protocol:

Three dentinal carious lesions will be chosen in this study and will be in the same patient. The lesions will be classified using the International Caries Detection and Assessment System (ICDAS-II). after air-drying the teeth using a triplex syringe ICDAS-II scores of the lesions will be obtained. The chosen sites will be recorded as: Code 4, non-cavitated Lesion extending into dentine seen as an undermining shadow; code 5, small cavitated lesion with visible dentine: less than 50 % of surface; code 6, large cavitated lesion with visible dentine: more than 50 % of surface. In all cases, dentine lesions were soft and wet indicating an active lesion.

Using local anaesthesia and rubber dam, the operative field will disinfected with 1% hypochlorite,and the dentine lesions should be exposed with a high-speed diamond bur by removing covering enamel.

Before the excavation dentine samples are collected for baseline bacteriological assessment . Excavation will be carried out using new slow speed round burs and hand excavators. Special consideration will be given to avoid pulpal exposures and over excavation. In order to avoid this, hand excavators will be used for the final excavation stage.

II.3.b Clinical assessment:

The excavation end point of one cavity will be determined using visual tactile method. The two other cavities will be inspected with fluorescent camera or caries detector dye (CDD) methods to determine excavation endpoint respectively. After excavation, dentine samples from the three cavities will be collected using a sterile excavator for the bacteriological assessment.

II.3.c Assessment of Outcome:

Samples of carious and sound dentine will be collected with sterile excavators after caries removal in the three groups. The dentine samples will be transferred to sterile box containing a thioglycollate medium used as a carrier, then this sterile box will be kept in an ice box and taken to the microbiology laboratory for processing, within an hour, by another examiner who do not know the type of technique used for the inspection after the caries excavation. Dentin sample weight will be calculated by measuring the difference between the weight of the whole set (sterilized bottle, transporting medium, collected dentine) and the previously determined weight of the set without dentin. The number of bacteria obtained for a given amount of dentin will be used to estimate the number of bacteria present in 1 mg dentin (CFU/mg).

II.4. Participant timeline:

All procedures will be carried out at the same visit.

II.5. Sample size calculation:

The aim of this study will be conducted to assess the reliability of the fluorescence camera and caries detection dye versus visual tactile method in caries excavation using bacteriological assessment method. Based on the previous paper by Stroll et al.,2015 ,area under the curve for fluorescent camera using bacterial count as reference was 0.75. Using power 80% and 5% significance level, 20 cavities is needed in each group the sample size was calculated by PASS 2008.

II.6. Recruitment:

Patients will be recruited from outpatient clinic of Conservative Dentistry Department in Faculty of Oral and Dental Medicine, Cairo University; from which eligible patients will be recruited to fulfil the eligibility criteria according to participant timeline.

II.6.a. Recruitment Strategy:

The patients will be subjected to full examination and diagnosis using dental charts. Once the patients that are potentially eligible for this study are identified, they will be contacted by the researcher who will explain the study and ascertains the patient's interest. If interested, more detailed evaluations and preparations are made.

II.7. Randomization and assignment of interventions:

II.7.a. Allocation sequence generation:

The allocation sequence will be generated using (www.randomization.com).

II.7.b. Allocation concealment mechanism:

Each recruited patient will be given a number according to order of recruitment following the sequence of the randomly generated numbers, then the operator will start the first tooth to be excavated, then will choose between three opaque sealed envelopes (two envelope for the intervention and the other is for the control). envelopes will be allocated by a participant who will not be involved in any of the phases of the clinical trial. The tooth to which interventions or control is assigned to will be recorded and all records of all patients will be kept with the main supervisor

II.7.c. Implementation:

A participant will generate the random allocation sequence. The researcher will enroll the patients but an unbiased participant will assign the intervention/Control to respective teeth.

II.8. Data collection methods:

*Baseline data collection:

For every patient medical history, dental history and examination charts will be filled by the operator.

*Outcome data collection:

The results were converted table to facilitate the description of the results. The microbiological analysis was performed blindly in relation to the caries removal method.

II.9.Data management:

the data will be entered and stored on a personal computer. Double data entry will be saved on an external hard disc to prevent loss of data.

II.10. Statistical methods

Data will be analyzed using IBM SPSS advanced statistics (Statistical Package for Social Sciences). Numerical data will be described as mean and standard deviation or median and range. Data will be explored for normality using kolmogorov-smirnov test and Shapiro-Wilk test. Comparisons between 3 groups for normally distributed numeric variables will be done using the ANOVA while for non normally distributed numeric variables will be done by Kruskal Wallis test. A p-value less than or equal to 0.05 will be considered statistically significant. All tests will be two tailed.

II.11. Monitoring:

II.11.a. Data monitoring:

The main supervisor will monitor this study. His role is to monitor any risk of bias could be done from participants, operator or assessors. Also to monitor blinding of the assessors and patient safety, outstanding benefits or harms.

II.11.b. Harms:

The main supervisor should inform participants about the possible harms, if present. Participants are allowed to contact the operator at moment through telephone. In case of accidental pulp exposure during excavation , emergency access cavity and pulp extirpation will be done by the operator and then the patient will be referred to Endodontic Department clinic to complete the root canal treatment.

II.11.c. Auditing:

In the present trial, auditing will be done by the main and co-supervisors to assure quality of the research frequency procedures.

II.14. Ethics and dissemination

II.14.a. Research ethics approval:

Application forms for carrying out the clinical trial, checklist and informed consent of Research Ethics Committee (REC) Faculty of Oral and Dental Medicine, Cairo University will be retrieved and filled, then will be delivered for (REC) committee for approval.This is done to prevent any ethical problems during the study or any harm for any of the participants.

II.12.b. Protocol amendments:

If a new protocol will be used a protocol amendment will be submitted; containing a new copy of the new protocol and brief explanation about the differences between it and the previous protocols. If there is a change in the existing protocol that affect safety of subjects, investigation scope or scientific quality of the trial, an amendment containing a brief explanation about the change will be submitted. If a new author will be added to accomplish the study, an amendment including the investigator's data and qualifications to conduct the investigation will be submitted to prevent ghost authorship.

II.12.c. Consent:

The operator is responsible for admitting and signing the written consents during the enrolment day.

II.13. Confidentiality:

Name, personal data and pictures of the participants will not appear on the protocol form and will be maintained secured for 10 years after the trial. This is done for protection of participants' privacy and civil rights.

II.16. Declaration of interests:

There is no conflict of interest, no funding or material supplying from any parties.

II.14. Access to data:

Access to final data will be allowed to the operator ,the main and co-supervisors of the study who are not involved in assessment of the outcome.

II.15. Ancillary and post-trial care:

Patients will be followed up after the application after 3, 6 months.

II.16. Dissemination policy:

Full protocol will be published online in www.clinicaltrials.gov to avoid repetition and to keep the integrity of the research work. Thesis will be discussed in front of judgment committee. The study will be published to report the results of this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with at least three carious lesions .
2. Males or Females.
3. Good oral hygiene.
4. Co-operative patients approving the trial.

Exclusion Criteria:

1. Pregnancy.
2. Systemic disease or severe medical complications.
3. Heavy smoking.
4. Xerostomia.
5. Lack of compliance.
6. Evidence of temporomandibular joint disorders.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-02-03 (Actual); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-03-30 (Estimated)

PRIMARY OUTCOMES:
bacterial count | an average of 1 year
  will be done by Digital colony counter, Agar diffusion test

CONTACTS AND LOCATIONS:
Overall Officials: mohamed riad farid, PHD, Study Director — Professor of Conservative Dentistry, Cairo university; Rasha Ra'faat Abdel Aziz, PHD, Study Chair — Lecturer of Conservative Dentistry, Cairo university
Locations (1):
- Mohamed Mohamed sabry Mohamed, Cairo, Nasr City, Egypt

IPD SHARING:
Plan to Share IPD: Yes
publishing the data at egyptian dental journal

REFERENCES:
- [Background] Stoll R, Urban-Klein B, Giacomin P, Loukas A, Jablonski-Momeni A. In vivo assessment of caries excavation with a fluorescence camera compared to direct bacteriological sampling and quantitative analysis using flow cytometry. Lasers Med Sci. 2015 Feb;30(2):843-9. doi: 10.1007/s10103-013-1459-2. Epub 2013 Oct 19. PMID 24142047